CLINICAL TRIAL: NCT04278651
Title: Early Antenatal Support for Iron Deficiency Anemia: A Randomized Controlled Trial of Early Initiation of Intravenous Versus Oral Iron Therapy for Treatment of Iron Deficiency Anemia in Pregnancy
Brief Title: Early Antenatal Support for Iron Deficiency Anemia
Acronym: EASI-A
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Auerbach Hematology and Oncology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19G.929
Record Dates: First submitted 2020-02-04; First posted 2020-02-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy Related; Anemia, Iron Deficiency; Anemia of Pregnancy
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral Iron (Active Comparator): 325mg oral iron (ferrous sulfate) twice daily
  Interventions: Drug: Ferrous Sulfate
- Intravenous Iron (Experimental): 510mg ferumoxytol intravenous infusion for two doses total; second dose 3-8 days after first dose.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — 510mg infusion x 2 doses 3-8 days apart
  Arms: Intravenous Iron
Drug: Ferrous Sulfate — 325mg oral twice daily
  Arms: Oral Iron

SUMMARY:
This is a randomized, controlled multi-site trial of iron therapy in pregnancy. The purpose of this research is to see if second trimester initiation of intravenous (IV) iron therapy is better than oral iron therapy for treatment of anemia in pregnancy by improving blood count, quality of life and reducing side effects.

DETAILED DESCRIPTION:
Pregnant singletons diagnosed with iron deficiency anemia will be enrolled between 14-24 weeks and will be randomized 1:1 to either a course of ferumoxytol (510mg x 2 doses 3-8 days apart) or oral iron (325mg) twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation
* Gestational age <24 weeks
* Baseline Hb ≥9.0 and <11.0 with evidence of iron deficiency anemia

Iron deficiency anemia diagnosed (at any point in patient history) by:

* Hb<11.0
* Ferritin<30 and/or total iron saturation <20

Exclusion Criteria:

* Sickle cell Disease (NOT sickle cell trait)
* Evidence of acute anemia requiring transfusion or IV iron therapy
* Major congenital or chromosomal anomaly
* Previous use of IV iron in this pregnancy
* Severe cardiac, renal, or liver disease
* Autoimmune disease (ie Systemic Lupus Erythematosus (SLE)
* Allergy or contraindication to either study drug
* History of medication allergy, reaction to IV infusion, or reaction to Feraheme or other IV iron products

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin | 90 days
  Change in hemoglboin at day 90 following treatment initiation

SECONDARY OUTCOMES:
Anemia resolution | 90 days
  Percent of participants in each group with Hb>=11.0 at day 90
Anemia at Delivery | 9 months
  Percent of participants in each group with Hb>=11.0 at delivery
Need for additional therapy | 9 months
  Percent of participants in each group requiring additional therapy for iron deficiency anemia after 28 weeks
Quality of life scale | 30, 60, 90 days
  Linear Analogue Scale Assessment
Adherence | 90 days
  adherence to assigned group. Measured by what % of IV infusions completed of the two required in IV iron group, and for oral iron group, what %pills taken/prescribed based on pill counts
Need for post partum transfusion | 9 months
  Incidence of transfusion after delivery/post partum
Neonatal outcomes: cord blood iron indices | 9 months
  Hb, ferritin, total iron saturation
Neonatal outcomes: birth weight | 9 months
  birth weight (grams)
Neonatal outcomes gestational age of delivery (weeks) | 9 months
  gestational age of delivery (weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of planned primary and secondary analysis, IPD data may be available on request with completion of appropriate data sharing agreements
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 1 year after publication of study results
Access Criteria: After completion of planned primary and secondary analysis, IPD data may be available on request with completion of appropriate data sharing agreements